CLINICAL TRIAL: NCT04714216
Title: Automated Insulin Delivery for INpatients With DysGlycemia (AIDING) Feasibility Study
Brief Title: Automated Insulin Delivery for INpatients With DysGlycemia (AIDING) Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Insulet Corporation (Industry); Jaeb Center for Health Research (Other)
Responsible Party: Principal Investigator, Francisco Pasquel, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001835
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus
Keywords: Automated insulin delivery; Hybrid closed-loop system; Inpatient insulin therapy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hybrid closed-loop (HCL) automated insulin delivery (AID) (Experimental): Hybrid closed-loop (HCL) automated insulin delivery (AID) using the Omnipod 5/Horizon HCL system with remote monitoring and device operation capabilities will be deployed to hospitalized patients admitted to the general medical/surgical floor with diabetes (type 1 or type 2) requiring insulin therapy.
  Interventions: Device: The Omnipod 5/Horizon HCL system

INTERVENTIONS:
Device: The Omnipod 5/Horizon HCL system — The Omnipod 5/Horizon HCL system, consists of a disposable insulin infusion pump (or "pod"), a built-in model predictive control (MPC) insulin dosing algorithm, and a remote Personal Diabetes Manager (PDM) interface, that interact with a Dexcom G6 continuous glucose monitor (CGM) to automatically control insulin delivery based upon real-time glucose values. The PDM component also enables remote interaction with the system, including glucose monitoring as well as insulin dosing management and adjustments.

SUMMARY:
This single-arm stepwise feasibility study will test initial deployment of hybrid closed-loop (HCL) automated insulin delivery (AID) using the Omnipod 5/Horizon HCL system with remote monitoring and device operation capabilities to hospitalized patients admitted to the general medical/surgical floor with diabetes (type 1 or type 2) requiring insulin therapy.

DETAILED DESCRIPTION:
This single-arm stepwise feasibility study will test initial deployment of hybrid closed-loop (HCL) automated insulin delivery (AID) using the Omnipod 5/Horizon HCL system with remote monitoring and device operation capabilities to hospitalized patients admitted to the general medical/surgical floor with diabetes (type 1 or type 2) requiring insulin therapy. All enrolled participants will be placed on HCL insulin therapy for 10 days or until hospital discharge (if less than 10 days) to determine functional operability of the system and its effect on glycemic control in the hospital setting. This study will generate preliminary data to inform the design of a large multi-institution randomized controlled trial to assess superiority of HCL compared to standard inpatient insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with insulin-treated T1 or Type 2 diabetes mellitus (T2DM) admitted to general (non-intensive care) medical-surgical hospital service requiring inpatient insulin therapy.

Exclusion Criteria:

* Patients admitted the ICU or anticipated to require ICU transfer
* Anticipated length of hospital stay <48 hours.
* Evidence of hyperglycemic crises (diabetic ketoacidosis or hyperosmolar hyperglycemic state) at enrollment
* Severely impaired renal function (eGFR < 30 ml/min/1.73m2) or clinically significant liver failure
* Severe anemia with hemoglobin <7 g/dL
* Evidence of hemodynamic instability
* Hypoxia (SpO2 <95% on supplemental oxygen)
* Pre-admission or inpatient total daily insulin dose >100 units
* Mental condition rendering the participant unable to consent or answer questionnaires
* Pregnant or breast feeding at time of enrollment
* Unable or unwilling to use rapid-acting insulin analogs (Humalog, Admelog, Novolog or Apidra) during the study
* Use of hydroxyurea or high-dose ascorbic acid (>1g/day)
* Coronavirus Disease 2019 (COVID-19) infection or person under investigation (PUI) on isolation precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Pasquel, M.D., M.P.H, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Grady Health System (non-CRN), Atlanta, Georgia
  - University of Virginia School of Medicine, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Health System in Atlanta, Georgia, Stanford University School of Medicine, California, and University of Virginia School of Medicine in Charlottesville, Virginia, USA. Participant enrollment began June 29, 2021 and all follow-up assessments were completed by August 11, 2022.
Groups:
- Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID): Hybrid closed-loop (HCL) automated insulin delivery (AID) using the Omnipod 5/Horizon HCL system with remote monitoring and device operation capabilities was deployed to hospitalized patients admitted to the general medical/surgical floor with diabetes (type 1 or type 2) requiring insulin therapy. The Omnipod 5/Horizon HCL system, consists of a disposable insulin infusion pump (or "pod"), a built-in model predictive control (MPC) insulin dosing algorithm, and a remote Personal Diabetes Manager (PDM) interface, that interact with a Dexcom G6 continuous glucose monitor (CGM) to automatically control insulin delivery based upon real-time glucose values. The PDM component also enables remote interaction with the system, including glucose monitoring as well as insulin dosing management and adjustments.
Period: Overall Study
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Started | 22
Completed | 18
Not Completed | 4
Not completed — Did not initiate AID due to CGM inaccuracies | 2
Not completed — Discharged prior to 48 hours of AID | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes participants who completed at least 48 hours of AID device use while hospitalized.
Groups:
- Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID): Hybrid closed-loop (HCL) automated insulin delivery (AID) using the Omnipod 5/Horizon HCL system with remote monitoring and device operation capabilities was deployed to hospitalized patients admitted to the general medical/surgical floor with diabetes (type 1 or type 2) requiring insulin therapy.
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 7
  White | 9
  More than one race | 1
  Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 31.2 [26.6 to 35.0]
Highest level of education [Count of Participants; unit: Participants]
  Less than high school diploma | 8
  High school completion or equivalent | 0
  Associate degree or some college | 6
  Bachelor's degree | 4
Annual household income [Count of Participants; unit: Participants] — Income measured in US Dollars (USD)
  Participants
    Less than $20,000 | 5
    $20,000-$49,999 | 3
    $50,000-$99,999 | 4
    ≥$100,000 | 2
    Declined to report | 4
Type of diabetes [Count of Participants; unit: Participants]
  Type 1 Diabetes | 2
  Type 2 Diabetes | 16
Duration of diabetes [Median (Inter-Quartile Range); unit: years] | 18 [10 to 20]
Most recent Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent of glycosylated hemoglobin] | 8.2 (1.4)
Modality of home insulin delivery [Count of Participants; unit: Participants]
  Injection | 15
  Insulin Pump | 0
  Not on insulin | 3
Primary reason for hospital admission [Count of Participants; unit: Participants]
  Cardiac | 6
  Respiratory | 2
  Infectious | 6
  Glycemic | 1
  Other | 3
Taking supraphysiologic doses of steroids [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent in HCL After CGM Sensor Meets Initial Validation Criteria
Description: The percentage of time spent in HCL after CGM sensor met initial validation criteria of sensor glucose value being within ±20% of point of care (POC) values (for glucose levels ≥70 mg/dL) or ±20 mg/dL for POC glucose values <70 mg/dL.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
percentage of time | 91 (11)

2. Primary Outcome: Percentage of Time Sensor Glucose is Within Target Glucose Range
Description: The percentage of time that the sensor glucose measurement is within the target glucose range of 70-180 mg/dL.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: Glycemic analysis using CGM metrics was prespecified in the study protocol to included participants with at least 48 hours of CGM data, thus, this analysis includes participants with at least 48 hours of CGM data. Although 18 participants used the device for 48 hours, only 16 had full CGM data for 48 hours.
Measure: Mean (Standard Deviation); unit: percentage of time in range (TIR)
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
percentage of time in range (TIR) | 68 (16)

3. Secondary Outcome: Time From Enrollment to Start of HCL Therapy (After Initial CGM Validation)
Description: The time from enrollment to start of HCL therapy, after initial CGM validation, was recorded.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
hours | 0 [0 to 0]

4. Secondary Outcome: Percentage of Time With CGM Readings
Description: The percentage of time during study participation with CGM readings was calculated.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
percentage of time | 99 [97 to 100]

5. Secondary Outcome: Percentage of CGM Values Meeting Accuracy Criteria for Bolus/Correction Insulin Dosing
Description: The percentage of CGM values meeting accuracy criteria for bolus/correction insulin dosing was calculated.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: This analysis includes 18 participants exposed to the to devices (Patch-pump and CGM device) for 48 hours.
Measure: Mean (Standard Deviation); unit: percentage of CGM values
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
percentage of CGM values | 85 (14)

6. Secondary Outcome: Percentage of CGM Readings Within %15/15 of POC Readings and Within %20/20 of POC Readings With the Cut Point at 70 mg/dL
Description: The percentage of CGM values within 15% or 15 mg/dL (%15/15) and within 20% or 20 mg/dL (%20/20) of POC reference values for blood glucose, using a cut point at 70 mg/dL. The reference values are derived from a total of 597 paired CGM and reference capillary glucose values.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: This analysis includes 18 participants exposed to the to devices (Patch-pump and CGM device) for 48 hours.
Measure: Mean (Standard Deviation); unit: percentage of CGM values
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
percentage of CGM values
  %15/15 of POC readings count | 71 (19)
  %20/20 of POC readings count | 81 (15)

7. Secondary Outcome: Number of Hypoglycemic (<70 mg/dL) Episodes Per Patient
Description: The number of hypoglycemic (<70 mg/dL) episodes per patient.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: Glycemic analyses using CGM metrics were prespecified in the study protocol to included participants with 48 hours or more of CGM data, thus, this analysis includes participants with at least 48 hours of CGM data. Although 18 participants used the device for 48 hours, only 16 had full CGM data for 48 hours.
Measure: Median (Full Range); unit: episodes per patient
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
episodes per patient | 0 [0 to 2]

8. Secondary Outcome: Number of Hypoglycemic (<70 mg/dL) Episodes Per Patient-day
Description: The number of hypoglycemic (<70 mg/dL) episodes per patient-day in hospital.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: episodes per patient-day
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
episodes per patient-day | 0 [0 to 0.3]

9. Secondary Outcome: Number Clinically Important Hypoglycemic (<54 mg/dL) Episodes Per Patient
Description: The number clinically important hypoglycemic (<54 mg/dL) episodes per patient.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: episodes per patient
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
episodes per patient | 0 [0 to 2]

10. Secondary Outcome: Percent Time Below Range (TBR) of <70mg/dL
Description: The percent time below range (TBR), defined as blood glucose <70mg/dL.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time below range
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
percentage of time below range | 0.17 (0.3)

11. Secondary Outcome: Percent Time Below Range (TBR) of <54 mg/dL
Description: The percentage of time below range (TBR) of <54 mg/dL.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time below range
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
percentage of time below range | 0.06 (0.2)

12. Secondary Outcome: Percent Time Above Range (TAR) of >180 mg/dL
Description: The percentage of time above range (TAR) of >180 mg/dL.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time above range
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
percentage of time above range | 25 (11)

13. Secondary Outcome: Percent Time in Severe Hyperglycemia (>250 mg/dL)
Description: The percentage of time in severe hyperglycemia, defined as >250 mg/dL.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
percentage of time | 6.9 (7.0)

14. Secondary Outcome: Frequency of Setting Overall Adjustments for Clinically-important Hypoglycemia (<54 mg/dL)
Description: The frequency of setting adjustments across all participants for clinically-important hypoglycemia, defined as <54 mg/dL.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 3

15. Secondary Outcome: Frequency of Setting Adjustments for Clinically-important Hypoglycemia (<54 mg/dL) to Basal Rate
Description: The frequency of setting adjustments across all participants for clinically-important hypoglycemia (<54 mg/dL) to basal rate.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 0

16. Secondary Outcome: Frequency of Setting Adjustments for Clinically-important Hypoglycemia (<54 mg/dL) to Insulin Carb Ratio (ICR)
Description: The frequency of setting adjustments across all participants for clinically-important hypoglycemia (<54 mg/dL) to insulin carb ratio (ICR).
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 3

17. Secondary Outcome: Frequency of Setting Adjustments for Clinically-important Hypoglycemia (<54 mg/dL) to Insulin Sensitivity Factor (ISF)
Description: The frequency of setting adjustments across all participants for clinically-important hypoglycemia (<54 mg/dL) to insulin sensitivity factor (ISF).
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 0

18. Secondary Outcome: Frequency of Setting Overall Adjustments for Prolonged Hyperglycemia (>250 mg/dL for >1 Hour)
Description: The frequency of setting adjustments across all participants for prolonged hyperglycemia, defined as blood glucose >250 mg/dL for over one hour.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 6

19. Secondary Outcome: Frequency of Setting Adjustments for Prolonged Hyperglycemia (>250 mg/dL for >1 Hour) to Basal Rate
Description: The frequency of setting adjustments across all participants for prolonged hyperglycemia, defined as blood glucose >250 mg/dL for over one hour, to basal rate.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 6

20. Secondary Outcome: Frequency of Setting Adjustments for Prolonged Hyperglycemia (>250 mg/dL for >1 Hour) to ICR
Description: The frequency of setting adjustments across all participants for prolonged hyperglycemia, defined as >250 mg/dL for over one hour, to ICR.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 25

21. Secondary Outcome: Frequency of Setting Adjustments for Prolonged Hyperglycemia (>250 mg/dL for >1 Hour) to ISF
Description: The frequency of setting adjustments across all participants for prolonged hyperglycemia, defined as blood glucose >250 mg/dL for over one hour, to ISF.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: setting adjustments
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
setting adjustments | 14

22. Secondary Outcome: Total Daily Insulin (TDI)
Description: The total daily insulin (TDI) was calculated.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
units/day | 0.41 (0.21)

23. Secondary Outcome: Total Daily Basal Insulin (TBI)
Description: The total daily basal insulin (TBI) was calculated.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
units/day | 0.21 (0.12)

24. Secondary Outcome: Total Daily Bolus Meal/Correction
Description: The total daily bolus meal/correction was recorded
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
units/day | 0.23 (0.13)

25. Secondary Outcome: Number of Hypoglycemic Events That Required Assistance of Another Person
Description: The number of hypoglycemic events across all participants that required assistance of another person due to altered consciousness to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: hypoglycemic events
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
hypoglycemic events | 0

26. Secondary Outcome: Number of Diabetic Ketoacidosis Events
Description: The number of diabetic ketoacidosis (DKA) events across all participants.
Time Frame: Up to 10 days (or hospital discharge if before 10 days)
Measure: Number; unit: DKA events
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 18
DKA events | 0

27. Secondary Outcome: Patient Acceptability of HCL System
Description: To assesses acceptability of the HCL system participants responded to the statement "Overall, I liked using the Omnipod 5/Horizon system to treat my blood sugar in the hospital" with five (5) options to choose from: Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, and Strongly Disagree. The responses were not assigned a score, rather the number of participants for each response were examined.
Time Frame: At time of device discontinuation (up to 10 days of use or hospital discharge if before 10 days)
Population: This analysis includes participants who completed the patient survey. Two participants were discharged from the hospital prior to completing the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
Participants
  Strongly Agree | 8
  Agree | 8
  Neither Agree nor Disagree | 0
  Disagree | 0
  Strongly Disagree | 0

28. Secondary Outcome: Patient Perceptions of HCL System Use
Description: Participants were asked to provide their perceptions of the HCL system with four questions that were responded to with "Yes" or "No". Responses are assigned a score and a summary score is not calculated, rather the number of participants responding "Yes" or "No" to each of the individual questions is examined.
Time Frame: At time of device discontinuation (up to 10 days of use or hospital discharge if before 10 days)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
Number analyzed (Participants) | 16
Participants
  "If you have diabetes, would you want to use this system to manage your diabetes at home?": Yes | 15
  "If you have diabetes, would you want to use this system to manage your diabetes at home?": No | 1
  "Did you find the number of alarms burdensome?": Yes | 0
  "Did you find the number of alarms burdensome?": No | 16
  "Did you find the number of fingersticks burdensome?": Yes | 6
  "Did you find the number of fingersticks burdensome?": No | 10
  "Would you prefer to use only the Dexcom sensory without the pump (pod)?": Yes | 3
  "Would you prefer to use only the Dexcom sensory without the pump (pod)?": No | 13

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected during exposure to study device, from the time individuals gave consent to participate (up to 10 days of use or hospital discharge if before 10 days).
Arm/Group | Hybrid Closed-loop (HCL) Automated Insulin Delivery (AID)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT04714216/Prot_SAP_000.pdf